CLINICAL TRIAL: NCT01260155
Title: A Single-Center, Open-Label, Randomized, 3-Treatment Crossover Bioavailability Study of Single Oral Doses of E5501 Old Tablet Formulation Under Fasted Conditions and a New Tablet Formulation Under Fed and Fasted Conditions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-005
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — avatrombopag

ARMS (3):
- Treatment A Fasted (Experimental)
  Interventions: Drug: E5501
- Treatment B Fasted (Experimental)
  Interventions: Drug: E5501
- Treatment C Food Effect (Experimental)
  Interventions: Drug: E5501

INTERVENTIONS:
Drug: E5501 — Treatment A: 40 mg new tablet formulation (1 tablet) under fasted conditions
  Arms: Treatment A Fasted
Drug: E5501 — Treatment B: 20 mg old tablet formulation (2 tablets) under fasted conditions
  Arms: Treatment B Fasted
Drug: E5501 — Treatment C: 40 mg new tablet formulation administered with food
  Arms: Treatment C Food Effect

SUMMARY:
This study will be a single-center, open-label, randomized, 3-treatment crossover bioavailability study of single oral doses of E5501 old tablet formulation under fasted conditions and a new tablet formulation administered under fed and fasted conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult males and females (age 18-45 years)
* Body Mass Index (BMI) greater than or equal to 18 and less than or equal to 32 at the time of Screening
* All females must have a negative serum human beta-chorionic gonadotropin test result or negative urine pregnancy test result at Screening and Baseline. Females of child-bearing potential must use a medically acceptable method of contraception throughout the entire study period and for 30 days after study drug discontinuation. Postmenopausal women and women who have been surgically sterilized or are proven sterile are exempt from this requirement. All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
* Male subjects who are not abstinent or have not undergone a successful vasectomy, who are partners of women of child-bearing potential must use, or their partners must use, a highly effective,method of contraception starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study period and for 30 days after the last dose of study drug.
* Willing and able to comply with all aspects of the protocol
* Provide written informed consent

Exclusion Criteria:

* Standard selection criteria typically used in all protocols
* Clinically significant abnormal laboratory test results, including platelet count and electrolyte abnormalities at Screening and at each Baseline

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the bioavailability (BA) of E5501 in one 40 mg new tablet formulation relative to two 20 mg old tablet formulation. | 2 months

SECONDARY OUTCOMES:
To determine the effect of a high fat meal on the BA of E5501 in one 40 mg new tablet formulation | 2 months
To evaluate the safety of E5501 in healthy subjects. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Johnson, Study Director — Eisai Inc.
Locations (1):
- Celerion, Phoenix, Arizona, United States